CLINICAL TRIAL: NCT05463458
Title: Evaluation of Immunonutrition For Patients With Pneumonia in the Intensive Care Unit.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azza Bahaa El-Din Ali Mohamed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: nutrition in ICU
Record Dates: First submitted 2022-06-19; First posted 2022-07-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Nutrition Poor
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): included 51 patients who will receive Standard of nutrition Care (2.0 g/kg body weight/day(A I) Calories should be in range of 25-30 Kcal/kg body weight/day.
  Interventions: Other: nutrition
- case (Experimental): included 51 patients who will receive adjusted and calculated dose of omega-3 polyunsaturated fatty acids (PUFA) and anti-oxidants.
  Interventions: Other: nutrition

INTERVENTIONS:
Other: nutrition — Standard of nutrition Care plus adjusted and calculated dose of omega-3 polyunsaturated fatty acids (PUFA) anti-oxidants.

SUMMARY:
The aim of the work will be to assess the combined effect of enteral or parenteral nutrition enriched with immunonutrition on the outcome of critically ill patients with pneumonia in comparison with patients who received standard care of nutrition in intensive care unit.

DETAILED DESCRIPTION:
Pneumonia is defined as an infection process of the lung parenchyma, which results from the invasion and overgrowth of microorganisms, breaking down defences, and provoking intra-alveolar exudates. Patients with pneumonia become malnourished ,exhibit declining health and changes in weight loss, and impair respiratory muscle contractility. Adequate nutrition aids respiratory muscle function and immune defence mechanisms. Therefore, the major role of nutrition in pneumonia is reducing malnutrition that induces high mortality and morbidity and maintaining impaired respiratory muscle contractility.

Pulmonary failure is associated with increased catabolism and decreased gut absorption. If respiratory failure require mechanical ventilation or patient need non-invasive ventilation. The presence of an artificial airway prevents volitional nutrition intake, leading to an energy deficit, the underlying process leading to respiratory failure may induce protein catabolism, causing loss of diaphragmatic and intercostal muscle mass, impairing immunity, impairing wound healing, and increasing the risk for new infection. Nutrition support also protects patients by minimizing malnutrition and loss of lean body mass.

Immunonutrition refers to modulation of the immune system provided by specific interventions that modify dietary nutrients. Several specialized enteral and parenteral formulas with immunonutrients are currently available on the market. These primarily consist of a combination of antioxidant vitamins (eg, vitamin C, vitamin E, ß-carotene), trace elements (eg, selenium, zinc), essential amino acids (eg, glutamine, arginine)or essential fatty acids, such as omega-3 fatty acids (eg, eicosapentaenoic acid, docosahexaenoic acid), and Ƴ-linolenic acid.

ELIGIBILITY:
Inclusion Criteria:

* Patients ( >18 years) with pneumonia requiring ventilatory support either invasive mechanical ventilation or non-invasive ventilation and could be enterally or parenterally fed in the respiratory intensive care unit of Assiut University Hospitals.

A diagnosis of pneumonia will be made based on clinical data and laboratory investigation. Radiological confirmation of the diagnosis will be done.

Patients will assess using the simplified acute physiology score (SAPS II) system (4). Also we will use nutric score.

Exclusion Criteria:

* Age less than 18 years old.
* Patients with immunosuppressive and malignant tumours. .Patients with severe liver and kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Effect of immunonutrition on : - Duration of mechanical ventilation. | 14 days
  Effect of immunonutrition on :
  * Duration of mechanical ventilation.

SECONDARY OUTCOMES:
Effect of immunonutrition on : - Blood oxygenation (PaO2/FiO2 ratio). | 14 days
  Effect of immunonutrition on :
  - Blood oxygenation (PaO2/FiO2 ratio).